CLINICAL TRIAL: NCT03514862
Title: Mindfulness Resiliency Training Pilot for University of Miami Medical Personnel
Brief Title: Mindfulness Training for Medical Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, David Lee, PhD, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180138
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Burnout, Professional; Stress
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will participate in 4 weeks of the Mindfulness-Based Intervention (MBI) and then will be invited to continue to participate in 4 additional Mindfulness Booster Training.
  Interventions: Behavioral: Mindfulness Booster Training; Behavioral: Mindfulness-Based Intervention (MBI)
- Control (Active Comparator): Participants will participate in 4 weeks of the Mindfulness-Based Intervention (MBI) and then continue to Self-Practice for 4 weeks.
  Interventions: Behavioral: Mindfulness Booster Training; Behavioral: Self-Practice

INTERVENTIONS:
Behavioral: Mindfulness Booster Training — Four additional mindfulness booster sessions after the 4-week MBI program.
Behavioral: Mindfulness-Based Intervention (MBI) — MBI program is delivered once a week for 4 weeks, 90 minutes each preceded by a 90-minute orientation session. The training sessions will include discussion, and introduction and practice of mindfulness practices.
  Arms: Intervention
Behavioral: Self-Practice — 4 weeks of self-practice after the MBI training.
  Arms: Control

SUMMARY:
In this project, the investigators propose to evaluate the impact of a Mindfulness-Based Intervention (MBI) Program on the well-being of University of Miami (UM) clinicians and faculty/staff. If successfully implemented and proven to be effective, this training program may be disseminated to other interested medical personnel.

ELIGIBILITY:
Inclusion Criteria:

* Medical faculty, fellows, residents, and other allied healthcare providers at UM Miller School of Medicine and Jackson will be eligible for participation in the study.

Exclusion Criteria:

* Those not falling into inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Change in measure of stress | Baseline, 4-weeks, 3-months, 6-months
  Stress will be measured using the Perceived Stress Scale, a short-form 4 item scale with a range of 0 to 16, with higher scores representing greater stress. Baseline responses will be compared to 4-week assessment responses of the control and intervention groups. Results between the control and intervention groups will be compared for statistical significance.

SECONDARY OUTCOMES:
Change in measure of burnout | Baseline, 4-weeks, 3-months, 6-months
  Burnout is measured using the 19-item Copenhagen Burnout Inventory including subscales assessing personal burnout, work-related burnout and patient-related burnout. Scores range from 0 to 100. Total score on the scale is the average of the scores on the items with a higher mean representing greater burnout. Baseline responses will be compared to 4-week assessment responses of the control and intervention groups. Results between the control and intervention groups will be compared for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: David J Lee, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No